CLINICAL TRIAL: NCT00004549
Title: MRI Detection of Vascular Inflammation in Patients Undergoing Peripheral Angioplasty
Brief Title: Magnetic Resonance Imaging to Detect Blood Vessel Inflammation in Patients Undergoing Peripheral Balloon Angioplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 000065; 00-H-0065
Record Dates: First submitted 2000-02-03; First posted 2000-02-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-01

CONDITIONS: Atherosclerosis; Peripheral Vascular Disease
Keywords: Atherosclerosis; Endothelium; Peripheral Vascular Disease; Markers of Inflammation; Claudication
MeSH Terms: conditions — Atherosclerosis; Peripheral Vascular Diseases; Intermittent Claudication | interventions — Magnetic Resonance Spectroscopy

INTERVENTIONS:
Procedure: Magnetic resonance imaging

SUMMARY:
This study will examine the use of magnetic resonance imaging (MRI) in detecting blood vessel inflammation. The results of this study may later be applied to diagnosing inflammation of arteries in patients with atherosclerosis, predicting disease progression in these patients, and guiding therapy.

Patients with peripheral artery disease (for example, blockage of a leg artery) undergoing balloon angioplasty at Suburban Hospital in Bethesda, Maryland, may be eligible to participate in this study. Because this procedure, which opens blocked arteries, can cause inflammation in the vessel wall, it affords an opportunity for studying MRI detection of such inflammation.

Study candidates will be screened with a medical history and physical examination. Participants will have a MRI scan and blood drawn at Suburban Hospital before the angioplasty and again either 1 to 3 days or 2 weeks after the procedure. Before the MRI scan is begun, a catheter (a thin plastic tube) is inserted in an arm vein and 90 milliliters (about 3 ounces) of blood is drawn. The patient then lies on a table that slides into the MRI scanner-a large donut-shaped machine with a magnetic field. A flexible, padded sensor called an MRI coil is placed over the area to be imaged; this device is used to improve the quality of the pictures. During the scan a contrast material called gadolinium is injected through the catheter. Gadolinium brightens the image of the blood vessels. The procedure lasts up to 2 hours.

DETAILED DESCRIPTION:
In this pilot study high resolution Magnetic Resonance Imaging (MRI) will be used to study 20 patients scheduled to undergo peripheral angioplasty in order to determine the MRI characteristics of acute and chronic vascular inflammation. The vascular territories to be angioplastied will be imaged in 20 patients with peripheral vascular disease prior to angioplasty. Patients will then be randomly assigned for imaging at 24-72 hours (10 patients) or imaging at 2-4 weeks (10 patients) post-angioplasty. Analysis will focus on paired comparisons between pre- and post-angioplasty data within each group. This study should provide data that can be applied to other research protocols designed to image inflammation associated with vascular injury and atherosclerosis.

ELIGIBILITY:
Must have clinically significant peripheral arterial disease and be referred from their physician for peripheral vascular angioplasty in the Suburban Hospital Radiology department.

Must be capable of giving informed consent.

Must be at least 18 years of age.

Must not have a history of severe claustrophobia.

Must not have a history of involuntary motion disorder.

Must not have a serum creatinine level greater than 2.0 mg/dL.

Must not have cardiac pacemaker or implantable defibrillator, aneurysm clip, neural stimulator (e.g. TENS-Unit), any type of ear implant, or metal in the eye (e.g. from machining).

Must not have systemic inflammatory disorder (e.g. systemic lupus erythematosus, rheumatoid arthritis, polyarteritis nodosa, Reiter's Syndrome).

Must not have the placement of a metal stent in the region to be imaged at the time of angioplasty.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2000-01; Study Completion 2002-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Libby P. Molecular bases of the acute coronary syndromes. Circulation. 1995 Jun 1;91(11):2844-50. doi: 10.1161/01.cir.91.11.2844. No abstract available. PMID 7758192
- [Background] Munro JM, Cotran RS. The pathogenesis of atherosclerosis: atherogenesis and inflammation. Lab Invest. 1988 Mar;58(3):249-61. PMID 3279259
- [Background] Navab M, Fogelman AM, Berliner JA, Territo MC, Demer LL, Frank JS, Watson AD, Edwards PA, Lusis AJ. Pathogenesis of atherosclerosis. Am J Cardiol. 1995 Sep 28;76(9):18C-23C. doi: 10.1016/s0002-9149(99)80466-4. PMID 7572682